CLINICAL TRIAL: NCT06975462
Title: SHR-A1811 Combined With Radiotherapy in HER2-positive and HER2-low Breast Cancer Brain Metastases: a Prospective，Sigle-arm，Phase II Study
Brief Title: A Phase II Study of SHR-A1811 Combined With Radiotherapy in HER2-positive and HER2-low Breast Cancer Brain Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UH-SHR A1811 and radiotherapy
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Metastatic
Keywords: breast cancer; barin metastases
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811+radiotherapy (Experimental): SHR-A1811:4.8mg/kg radiotherapy:800cGY*5
  Interventions: Combination Product: SHR-A1811 and radiotherapy

INTERVENTIONS:
Combination Product: SHR-A1811 and radiotherapy — SHR-A1811:4.8mg/kg radiotherapy: 800cGY*5

SUMMARY:
A prospective, single-arm study to explore the efficacy and safety of SHR-A1811 combined with radiotherapy in patients with HER2-positive or HER2-low brain metastases

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed HER2 positive (IHC 3+ or IHC 2+/FISH+)or HER2-low(IHC1+ or 2+/FISH-) advanced breast cancer
2. Age>18 years.
3. newly diagnosed Brain metastases confirmed by enhanced brain MRI. Metastases number less than 6.
4. No more than four lines of previous advanced therapy
5. Life expectancy of more than 3 months
6. There were no known or suspected leptomeningeal brain metastases
7. The interval from previous therapy was more than 2 weeks, and acute toxicity from previous therapy had to resolve to grade 1 or less
8. The use of mannitol, bevacizumab, or hormone therapy was allowed before enrollment, but the dose was stable for at least a week without the need for an increment
9. Screening laboratory values must meet the following criteria( and should be obtained within 28 days prior to registration):

Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L, Platelets≥ 90 x 109/L, Hemoglobin ≥ 90 g/L Aspartate aminotransferase/alanine aminotransferase (AST/ALT) ≤2.5 x ULN without liver metastasis,≤ 5 x ULN with liver metastases Serum BUN and creatinine ≤ 1.5 x Upper Limit of Normal (ULN) LVEF ≥ 50% QTcF < 480 ms INR≤1.5×ULN，APTT≤1.5×ULN 10.Signed the informed consent form prior to patient entry

Exclusion Criteria:

1. Leptomeningeal or hemorrhagic metastases
2. previously used T-dxd
3. Uncontrolled epilepsy
4. Severe or uncontrolled disease: severe cardiovascular disease, end-stage renal disease, severe hepatic disease, history of immunodeficiency, including HIV positive, active HBV/HCV or other acquired congenital immunodeficiency disease, or organ transplantation history, active infection, etc.
5. History of allergy to treatment regimens
6. Pregnancy or lactation period， women of child-bearing age who are unwilling to accept contraceptive measures.
7. Inability to complete enhanced MRI
8. Not suitable for inclusion for specific reasons judged by sponsor -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The objective response rate of intracranial（IC-ORR） | 2 years
  Proportion of participants with a complete response (CR) or partial response (PR) for intracranial tumors

SECONDARY OUTCOMES:
Intracranial CNS Progression Free Survival(IC-PFS) | 2 years
  Time from treatment until the first date of intracranial disease progression or death due any cause. For participants whose disease has not progressed at the time of the analysis, censoring will be performed using the date of the last valid disease assessment.
Progression Free Survival(PFS) | 2 years
  Time from treatment until the first date of intracranial or extracranial disease progression or death due any cause. For participants whose disease has not progressed at the time of the analysis, censoring will be performed using the date of the last valid disease assessment.
Overall survival(OS) | 3 years
  Time from the treatment until to the date of death, regardless of the cause of death
Adverse Events | 2 years
  Treatment-related adverse events were assessed and graded according to CTCAE v. 5.0

IPD SHARING:
Plan to Share IPD: No